CLINICAL TRIAL: NCT02203669
Title: The Use of Occupational/Physical Therapy to Reduce Upper Extremity Morbidity Post-Operative Bilateral Breast Reconstruction
Brief Title: Occupational/Physical Therapy to Reduce Morbidity Post-Operative Bilateral Breast Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never did begin
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OTPT2014
Record Dates: First submitted 2014-07-24; First posted 2014-07-30 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2014-07

CONDITIONS: Occupational/Physical Therapy; Post-operative Breast Reconstruction
Keywords: breast reconstruction; occupational therapy; physical therapy; upper extremity morbidity
MeSH Terms: interventions — Home Infusion Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Structured In-Office Therapy (Active Comparator): Structured In-Office Therapy: Study subjects will receive structured, therapist-supervised occupational/physical therapy twice per week for four (4) weeks. Each visit will last approximately sixty (60) minutes. Patients in this arm will receive therapy instruction by a certified occupational therapist on upper extremity stretching, relaxation, cardio rehabilitation, and strength training. These patients will also receive exercise and stretching handouts to use at home between therapy visits. Will complete the DASH at week 1 and week 4.
  Interventions: Other: Structured In-Office Therapy
- No therapy (No Intervention): Study subjects in this arm will not receive post-operative occupational /physical therapy. Will complete the DASH at week 1 and week 4.
- Home Therapy (Active Comparator): Home Therapy: Study subjects will receive a handout of exercises adapted for post-operative breast reconstruction patients along with an instructional handout for stretching complied by a certified occupational therapist to complete independently at home for four (4) weeks. Will complete the DASH at week 1 and week 4.
  Interventions: Other: Home therapy

INTERVENTIONS:
Other: Home therapy — Study subjects complete home therapy independently for four (4) weeks based on handouts of exercises adapted for post-operative breast reconstruction patients along with an instructional handout for stretching complied by a certified occupational therapist.
  Arms: Home Therapy
Other: Structured In-Office Therapy — Study subjects will participate in Structured In-Office Therapy twice a week for four (4) weeks. Each visit will last approximately sixty (60) minutes. Subjects will receive therapy instruction by a certified occupational therapist on upper extremity stretching, relaxation, cardio rehabilitation, and strength training. These subjects will also receive exercise and stretching handouts to use at home between therapy visits.
  Arms: Structured In-Office Therapy

SUMMARY:
The purpose of this study is to demonstrate the benefits of a structured occupational/physical therapy program on upper extremity morbidity for patients who have received bilateral breast reconstruction in comparison to a home therapy program and no post-operative therapy.

Hypothesis: Patients who engage in therapist-supervised occupational therapy following bilateral breast reconstruction have less upper extremity morbidity than those patients who complete a home therapy program or no therapy program.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Women who have had bilateral breast reconstruction
* All cancer stages will be included
* Physically and mentally able to participate in the study within the required time-frame
* Able to voluntarily give full informed consent to participate in the study

Exclusion Criteria:

* Women undergoing unilateral breast reconstruction
* Unable to provide informed consent in English
* Physically unable to engage in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change in DASH: Disabilities of the Arm, Shoulder and Hand score | Week 1 and Week 4
  A change in DASH score will be calculated. The DASH: Disabilities of the Arm, Shoulder, and Hand (Appendix D) questionnaire will be utilized to measure physical function and symptoms of the upper limbs. The DASH consists of 30-items to be self-reported by the patient: physical function twenty-one (21) items, pain symptoms five (5) items, and emotional and social function four (4) items. The result of the DASH is a numerical disability score ranging from zero to one hundred (0-100), with zero (0) being no disability and one hundred (100) being the most severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Brzezienski, MD, Principal Investigator — The University of Tennessee
Locations (1):
- The Plastic Surgery Group, P.C., Chattanooga, Tennessee, United States